CLINICAL TRIAL: NCT07401901
Title: Evaluation of the Safety and Effectiveness of the Novel Medtronic Experimental Automated Insulin Delivery System (NMX8) in Adults Living With Type 1 Diabetes
Acronym: ELEVATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP353
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Automated insulin delivery (AID); Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Helping Behavior; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment arm (NMX8 system) (Experimental): Subjects randomized to the Treatment group will use the MiniMed NMX8 system
  Interventions: Device: NMX8 System - Treatment arm
- Control arm (AID Therapy) (Active Comparator): Subjects randomized to the Control group will continue to use their current AID therapy during the study phase for 6-month. During the continuation phase, subjects in the Control group will use the NMX8 system for 3-month.
  Interventions: Device: AID Therapy; Device: NMX8 System - Control Arm

INTERVENTIONS:
Device: NMX8 System - Treatment arm — Subjects start using the NMX8 system after the run-in phase and continue through both study (6-month) and continuation phases (3-month).
  Arms: Treatment arm (NMX8 system)
Device: AID Therapy — Subjects will continue to use their current AID therapy during the study phase (6-month).
  Arms: Control arm (AID Therapy)
Device: NMX8 System - Control Arm — Subjects start using the NMX8 system during the continuation phases (3-month).
  Arms: Control arm (AID Therapy)

SUMMARY:
The purpose of the study is to evaluate the safety and the effectiveness of the Novel Medtronic Experimental Automated Insulin Delivery system, named MiniMed NMX8 system (referred also to as NMX8 system), in comparison with other commercially available AID systems (Automated insulin delivery) in adult patients with Type 1 diabetes not achieving target clinical outcomes.

DETAILED DESCRIPTION:
ELEVATE is a pre-market, interventional, prospective, open-label, multi-center, randomized controlled study that consists of three phases: run-in, study and continuation phase.

Run-in: the purpose of this phase is to collect 3 weeks of blinded Continuous Glucose Monitoring (CGM) data while subjects are on their current therapy (baseline assessment). All subjects will use an additional blinded Simplera Sensor to collect blinded CGM data.

Study Phase: during the 6-month of study phase subjects will either start using the NMX8 system (Treatment arm) or will continue to use their current AID therapy (Control arm). Subjects in the Control arm will undergo 3 weeks of blinded CGM data collection via Simplera Sensor at 3 and 6 months.

Continuation Phase: during the 3-month of continuation phase all subjects will use the NMX8 system.

Approximately 230 subjects will be enrolled in the study up to approximately 22 investigational centers in EMEA.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged ≥ 18 years old at time of screening.
2. Has a clinical diagnosis of Type 1 diabetes for ≥6 months prior to screening as determined via medical record by an individual qualified to make a medical diagnosis.
3. Is on commercially approved AID therapy (e.g. MiniMed 780G, Control IQ, OmniPod 5, CamAPS FX) for at least 3 months before screening.
4. Has a glycosylated hemoglobin (HbA1c) above 7% (53 mmol/mol), therefore is not achieving therapy goal, at time of screening visit (as processed by a Central Lab).
5. Must have a minimum daily insulin requirement (Total Daily Dose) of ≥ 6 units and a maximum of 250 units.
6. Has shown good compliance (≥80%) with sensor wear over the previous month prior to enrollment (based on sensor usage from the download summary report over the 30 days prior to enrollment).
7. Is willing to switch to an approved insulin per insulin pump labeling.
8. Is willing to participate in all training sessions as directed by study staff.
9. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol.
10. Subject is willing and able to provide written informed consent.

Exclusion Criteria:

1. Has untreated Addison's disease, thyroid disorder, growth hormone deficiency, hypopituitarism or definite gastroparesis, per investigator judgment.
2. Is using any anti-diabetic medication other than insulin at the time of the screening or plan on using during the study (e.g., pramlintide, DPP-4 inhibitor, GLP-1 and GIP agonists/mimetics, metformin, SGLT2 inhibitors).
3. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take chronically any oral, injectable, or IV glucocorticoids during the course of the study.
4. Has had renal failure defined by creatinine clearance <30 ml/min, as assessed by local lab test ≤ 6 months before screening or performed at screening at local lab, as defined by the creatinine-based Cockcroft, CKD-EPI or MDRD equations.
5. Has any unresolved adverse skin conditions in the area of sensor placement (e.g. psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
6. Has active or severe retinopathy in the last 6 months before the screening.
7. Has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
8. Has a positive pregnancy test at screening or plan to become pregnant during the course of the study or is breast feeding at the time of the enrollment.
9. History of 2 or more DKA events in the last 3 months before screening.
10. Is on "DIY" therapy at the time of the screening or at least 3 months before the screening.
11. Is planning to change AID therapy during the course of the study. Note: subjects randomized in the Control Arm should remain on their current therapy during the course of the study.
12. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrollment into this study, as per investigator judgment.
13. Is currently abusing illicit drugs, marijuana, alcohol or prescription drugs (other than nicotine), per investigator judgment.
14. Is part of the research staff involved with the study.
15. Is legally incompetent, illiterate or vulnerable person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2027-11-04 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | End of 6-month study phase
  The between-treatment difference (control arm using AID system vs treatment arm using the NMX8 system) in the percentage of time that the sensor glucose (SG) measurement is in the target range, 70 to 180 mg/dL (3.9-10.0 mmol/L) at the end of the study phase .
  The endpoint will be assessed for non-inferiority.

SECONDARY OUTCOMES:
Secondary Endpoint 1 | End of 6-month study phase.
  The between-treatment difference (control arm using AID system vs treatment arm using the NMX8 system) in HbA1c (%) at the end of the study phase.
  The endpoint will be assessed for non-inferiority.
Secondary Endpoint 2 | End of 6-month study phase.
  The between-treatment difference (control arm using AID system vs treatment arm using the NMX8 system) in HbA1c (%) at the end of the study phase.
  The endpoint will be assessed for superiority.
Secondary Endpoints 3 | End of 6-month study phase.
  The between-treatment difference (control arm using AID system vs treatment arm using the NMX8 system) in the percentage of time spent in target range 70 to 180 mg/dL (3.9-10.0 mmol/L) at the end of the study phase.
  The Endpoint will be assessed for superiority.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ohad Cohen, MD, Study Chair — Medtronic Diabetes
Locations (20):
- France (5):
  - Centre Hospitalier Universitaire de Caen, Caen
  - Hôpital Michallon - CHU Grenoble, Grenoble
  - Hospices Civils de Lyon (DIAB-e CARE), Lyon
  - CHU de Nîmes - Hôpital Universitaire Caremeau, Nîmes
  - Hopital Lariboisiere & Fernand-Widal, Paris
- Germany (3):
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bad Oeynhausen
  - Zentrum für digitale Diabetologie Hamburg, Hamburg
  - Die Praxisgemeinschaft für Endokrinologie und Diabetes, Rostock
- Italy (4):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli - Università Cattolica del Sacro Cuore, Roma
- Netherlands (3):
  - ZGT Almelo, Almelo
  - Diabates Center Amsterdam, Amsterdam
  - Maastricht University Medical Center (UMC), Maastricht
- Spain (2):
  - Hospital Universitari Clínic de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
- United Kingdom (3):
  - University Hospitals of Derby and Burton NHS Foundation Trust - Florence Nightingale Community Hospital, Derby
  - Leicester General Hospital, Leicester
  - Manchester University NHS Foundation Trust - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No